CLINICAL TRIAL: NCT01967277
Title: A Novel Approach to Treating Androgenetic Alopecia in Females With Low Level Laser Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capillus, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: USC650
Record Dates: First submitted 2013-10-18; First posted 2013-10-22 (Estimated); Results first posted 2015-05-06 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Incandescent red light source (Placebo Comparator): A red, incandescent light source replaces all laser output. The treatment sessions are self-administered at home, every other day, for 16 weeks.
  Interventions: Device: Incandescent red light source.
- Handi-Dome Laser (Active Comparator): Study subjects self-administer actual laser treatments, at home, every other day, for 16 weeks.
  Interventions: Device: Handi-Dome Laser

INTERVENTIONS:
Device: Handi-Dome Laser — One, 30 minute treatment, every other day for 16 weeks.
  Arms: Handi-Dome Laser
Device: Incandescent red light source. — One, 30 minute treatment, every other day for 16 weeks.
  Arms: Incandescent red light source

SUMMARY:
This study will acquire data on hair growth of the head that is the result of treatment with a non-heat generating, laser product. This data will come from counting of terminal hairs before treatment begins and after treatment is completed. The treatment regime is every other day for 16 weeks.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy of Low Level Laser Therapy product that is configured in the novel design of a baseball cap, for promoting hair growth in females diagnosed with genetic hair loss/female pattern hair loss.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of Androgenetic Alopecia / Female Pattern Hair Loss Fitzpatrick skin phototypes of I - IV Ludwig-Savin Hair Loss scale I - II In overall good health as determined by the physician investigator Active hair loss within the last 12 months Willingness to refrain from using all other hair growth products or treatments -

Exclusion Criteria:

Photosensitivity to the specific wavelength of light - 650 nanometers. Malignancy in the target treatment area Other forms of alopecia of the head Past medical history of a collagen-vascular disease, thyroid disease or other cutaneous or systemic disease that seriously affects the scalp.

In willingness to remove hair replacement products during the 16 weeks of therapy.

Using any medications deemed to inhibit hair growth as determined by the physician investigator.

-

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2014-03; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond R. Blanche, BA, Study Director — NST Consulting, LLC
Locations (2):
- United States (2):
  - Bodian Dermatology, Great Neck, New York
  - Center for Aesthetic Dermatology, Woodbury, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Incandescent Red Light Source: Placebo: A red, incandescent light source replaces all laser output. The treatment sessions are self-administered at home, every other day, for 16 weeks.
  Incandescent red light source.: One, 30 minute treatment, every other day for 16 weeks.
- Handi-Dome Laser: Active Device: Study subjects self-administer actual laser treatments, at home, every other day, for 16 weeks.
  Handi-Dome Laser: One, 30 minute treatment, every other day for 16 weeks.
Period: Overall Study
Arm/Group | Incandescent Red Light Source | Handi-Dome Laser
Started | 22 | 22
Completed | 21 | 19
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Unrelated illness | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Incandescent Red Light Source | Handi-Dome Laser | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Median (Full Range); unit: years] | 49 [28 to 60] | 49.5 [28 to 58] | 49 [28 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 44
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Percentage Increase in Terminal Hair Counts From Pre-Treatment, Baseline for Active Test Subjects Over the Placebo Test Subjects.
Description: At baseline, a 25 mm area of treatment was trimmed of hair (to 3mm) at the vertex of the scalp and photographs were taken, terminal hairs were counted.
Time Frame: baseline and 17 weeks
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Incandescent Red Light Source | Handi-Dome Laser
Number analyzed (Participants) | 21 | 19
percent change | 12.48 (13.76) | 63.67 (50.9)
Statistical Analysis 1: Comparison: Incandescent Red Light Source vs Handi-Dome Laser; H0: µL ≤ µs Versus Ha: µL > µs; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

2. Primary Outcome: Absolute Increase in Terminal Hair Counts From Pre-Treatment, Baseline for Active Test Subjects Over the Placebo Test Subjects.
Description: as for outcome 1
Time Frame: baseline and 17 weeks
Measure: Mean (Standard Deviation); unit: terminal hairs
Arm/Group | Incandescent Red Light Source | Handi-Dome Laser
Number analyzed (Participants) | 21 | 19
terminal hairs
  Hair count, baseline | 216.9 (109.1) | 189.3 (85.8)
  Hair count, post treatment | 235.3 (105.8) | 268.3 (117.7)
  Hair count, difference | 18.5 (24.4) | 89.9 (63.3)

ADVERSE EVENTS:
Arm/Group | Incandescent Red Light Source | Handi-Dome Laser
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI may not disclose the results of the trial.